CLINICAL TRIAL: NCT07068984
Title: Assessing Lower Extremity Dynamic Stability in Middle-Aged and Elderly Patients With Patellofemoral Pain Using the Y-Balance Test: A Cross-Sectional Study
Brief Title: Assessing Lower Extremity Dynamic Stability in Middle-Aged and Elderly Patients With Patellofemoral Pain Using the Y-Balance Test
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022744
Record Dates: First submitted 2025-05-28; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: Y-balance; Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A total of 49 patients with PFPS and 21 healthy controls were enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Twenty-one healthy controls were enrolled: 2
  Interventions: Other: Differences between lower limb balances were assessed by the Y-Balance test
- A total of 49 patients with PFPS and 21 healthy controls were enrolled

INTERVENTIONS:
Other: Differences between lower limb balances were assessed by the Y-Balance test — The Y-Balance test was used to evaluate bilateral anterior difference, composite score, lateral and posterior balance, symmetry ratio and bilateral difference
  Groups: Twenty-one healthy controls were enrolled

SUMMARY:
Background: Patellofemoral pain syndrome (PFPS) is a common functional disorder of knee joint. Its etiology involves biomechanical abnormalities and dynamic stability defects. Most of the existing studies focus on young people, and the biomechanical characteristics and functional compensation mechanism of middle-aged and elderly patients are still unclear. The Y-Balance test is becoming an important tool in PFPS research because of its sensitivity to assess the dynamic balance ability of lower limbs. Objective: To analyze the functional characteristics of lower limbs of PFPS patients aged 40-60 by Y-Balance test, and to explore the differences between PFPS patients and healthy people, so as to provide evidence for clinical rehabilitation. Methods: A cross-sectional observational study was conducted in 49 PFPS patients and 21 healthy controls. Y-Balance test was used to evaluate bilateral forward difference, composite score, lateral and posterior balance, symmetry ratio and bilateral difference. SPSS 25.0 was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 60 years
* Clinically diagnosed with patellofemoral pain (PFP) with symptoms lasting ≥3 months
* No other serious lower extremity disorders
* No neurological diseases
* No history of recent lower extremity surgery (<12 months)
* No history of major lower extremity trauma
* Control group: Age- and sex-matched healthy volunteers without knee pain or lower limb dysfunction

Exclusion Criteria:

Acute inflammatory conditions Meniscus injury Knee ligament injury Intra-articular fracture Bone tumor Bone tuberculosis

Neurovascular injury including:

1. Stroke history
2. Parkinson's disease Subjective unwillingness to comply with testing Inability to complete Y-Balance Test

Serious systemic diseases affecting:

Cardiovascular system Hepatic function Renal function Hematological system

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: People with patellar pain
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Analysis of Y-balance characteristics of patellofemoral pain syndrome | Baseline
  Outcome Measure Title:Y-Balance Test (YBT) Reach Distance (cm) - Comparison between Patellofemoral Pain Syndrome (PFPS) Patients (Aged 40-60 Years) and Healthy Controls Outcome Measure Description:The Y-Balance Test (YBT) was used to assess dynamic balance function of the lower limbs in participants.
  Metrics Measured: The maximum reach distance (in centimeters, cm) achieved by participants in three directions (Anterior, Posteromedial, Posterolateral) during single-leg stance.
  Data Summary:The average maximum reach distance (cm) from three valid trials was calculated for each direction, separately for the left and right legs.
  Comparative Analysis: The average maximum reach distance (cm) in each direction for the left and right legs in the PFPS patient group (aged 40-60 years) were compared with the corresponding metrics in an age- and sex-matched group of healthy controls to analyze between-group differences.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zheng Z, Fan H, Hongjie H, Jianquan W. Deficits in dynamic stability revealed by the Y-Balance test in middle-aged and elderly adults with patellofemoral pain. J Orthop Surg Res. 2026 Jan 28. doi: 10.1186/s13018-026-06684-9. Online ahead of print. PMID 41593626